CLINICAL TRIAL: NCT06184100
Title: Feasibility and Acceptability of a Virtual Self-management Program - A Pilot Randomized Controlled Trial for Adolescents With Juvenile Idiopathic Arthritis
Brief Title: Virtual Self-Management Program for JIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The Hospital for Sick Children (Other); University of Toronto (Other); University of Alberta (Other); University of Manitoba (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VISTA-JIA
Record Dates: First submitted 2023-11-10; First posted 2023-12-28 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Virtual; Education; Clinical Trial; JIA; Self-management Program
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into an interventional or control group. The control group will be given the option to receive the intervention after post-test outcome measures are recorded.
Masking Description: The research team and all participants will be aware which arm they are enrolled in throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMP Program with Standard Care (Experimental): four 60-90 minute virtual educational sessions over 8 weeks with a group of 4-6 participants
  Interventions: Other: Virtual Self-Management Program (SMP)
- Standard Care Only (Active Comparator): Standard of care(no formal education program similar to SMP) and placed on 8-week waitlist for optional intervention.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Virtual Self-Management Program (SMP) — Four sessions, 60-90 minutes each, will be conducted over eight weeks with a group size of 4-6 participants via videoconferencing platforms such as Zoom or Microsoft Teams. Each session will include Power Point delivered presentations, interactive activities, and group discussions. This is a multifaceted program that includes JIA disease education, self-management strategies, and peer support.
  Arms: SMP Program with Standard Care
Other: No Intervention — No intervention. Participant only receives standard of care.
  Arms: Standard Care Only

SUMMARY:
The aim of this project is to conduct a pilot randomized controlled trial (RCT) to evaluate the feasibility and preliminary effectiveness of a virtual group based self-management program (SMP) in adolescents with JIA across different provinces compared to a wait-list control group receiving only standard of care.

Participants in the SMP group will partake in four 60-90 minute group sessions conducted over 8 weeks. The intervention is a multifaceted program that includes JIA disease education, self-management strategies, and peer support. Both the interventional and control group will be asked to complete baseline and post-test measures.

Participants in the control group will be offered the SMP after completion of the post-control outcome measures.

DETAILED DESCRIPTION:
A pilot RCT will be conducted to evaluate the feasibility and preliminary effectiveness comparing the SMP intervention group with a wait-list control group receiving usual care. A total of 100 participants with confirmed JIA (ages 12 to 17) will be recruited from five Canadian pediatric rheumatology centres of different provinces and randomized in a 1:1 ratio to the control or intervention groups. Adolescents in the intervention group will receive the virtual SMP program in addition to standard of care. The intervention is a multifaceted program that includes JIA disease education, self-management strategies, and peer support. Four 60-90- minute sessions will be conducted over eight weeks with a group size of 4-6 participants. Both groups will receive usual care. Participants in the control group will be offered the SMP after completion of the post-control outcome measure. If participants choose to enroll in the SMP, the participants will be asked to complete outcome measures a second time upon completion of the program.

The primary objective is feasibility outcome that will be measured as adherence with the SMP Program (defined as 80% completion). Other feasibility outcomes will include:

(A) recruitment and withdrawal rates (>80% recruitment rate and <80% withdrawal); (B) proportion of completed questionnaires (C) engagement and satisfaction with the SMP program as measured through a semi-structured virtual interview with the participants following involvement in the SMP; (D) intervention fidelity (consistent content and technology delivery).

The secondary objective on preliminary effectiveness includes completion of five validated and reliable patient-reported outcome measures at two-time points: perceived ability to manage JIA (self-management), pain interference, self-efficacy, health-related quality of life (HRQL) and transition readiness. These questionnaires will include:

(A) Medical Issues, Exercise, Pain, and Social Support Questionnaire (MEPS), (B) Children's Arthritis Self-Efficacy Scale (CASES), (C) Pediatric Quality of Life Inventory 3.0 Rheumatology - Teen Module (Peds QL, (D) PROMIS Pediatric Pain Interference Scale (PROMIS) and RACER (Readiness for Adult Care in Rheumatology). Descriptive statistical methods and non-parametric tests will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents between the ages of 12 and 17
2. Confirmed diagnosis within 2 years according to the International League of Associations for Rheumatology JIA classification criteria (2)
3. Followed in one of the pediatric rheumatology clinics participating in the RCT
4. Able to access the Internet on a computer
5. Willing and able to complete online measures

Exclusion Criteria:

1. Insufficient English reading and speaking skills
2. Untreated psychiatric or comorbid disorders or major cognitive impairments leading to inability to understand materials and participate in the SMP group activities.
3. Other chronic conditions such as other autoimmune disease, neurologic, orthopedics or other systems disorder (e.g. heart, kidney) that might influence outcome assessments
4. Past participation in the last year or participating in another peer-support or self-management program

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Program Adherence Rates (feasability) | 3 months
  The primary objective is feasibility outcome that will be measured as adherence with the SMP Program. This is defined as Proportion of completed questionnaires (defined as 80% when all measures are completed) at baseline and 8 weeks post-randomization in both groups along with recruitment and withdrawal rates. (>80% recruitment rate and <80% withdrawal)
Satisfaction of Program | 3 months
  Satisfaction with the SMP as measured through a semi-structured virtual interview with the participants following involvement in the SMP to capture participants' experience.
Intervention fidelity | 3 months
  We are looking at consistent content and technology delivery. This will be assessed by i) Observational checklists ii) qualitative analysis of recorded video sessions after 2, 4 and at completion of all sessions by each facilitator to ensure sessions are consistently delivered and as planned.

SECONDARY OUTCOMES:
Understanding of JIA | 3 months
  The medical issues, exercise, pain, and social-support [MEPS] questionnaire is a measure for perceived ability (e.g., knowledge, skill, behavior, attitudes, and self-efficacy) to manage JIA .
Understanding of Arthritis Self Efficacy | 3 months
  The Children's Arthritis Self-Efficacy Scale is a validated (e.g., concurrent validity, construct validity) and reliable (e.g., internal consistency) measure used for arthritis self-efficacy.
Quality of Life for Teens | 3 months
  The Pediatric Quality of Life Inventory 3.0 Rheumatology Teen Module is a validated (e.g. construct validity) and reliable (e.g., internal consistency) measure used for pediatric rheumatology specific health related quality of life in children aged 13-18
Physical Pain Level | 3 months
  The PROMIS Pediatric Pain Interference Scale is validated and reliable (e.g., internal consistency) measure for pain behavior in children aged 8-17
How Prepared the patient feels for Adult Care | 3 months
  Readiness for Adult Care in Rheumatology (RACER) questionnaire a reliable and validated instrument used to assess transition readiness in adolescents with JIA.

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth J, Birnie KA, Chomistek K, Santana M, Stinson JN, Adebiyi BO, Brooks J, Guzman J, Hellweg R, Lim LS, Rumsey D, Feldman BM, Tagseth J, Wilson J, Schmeling H. A Virtual Self-Management Intervention for Adolescents With Juvenile Idiopathic Arthritis: Protocol for the VISTA-JIA Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 27;14:e69539. doi: 10.2196/69539. PMID 40577780